CLINICAL TRIAL: NCT06344299
Title: Department of Hepato-Biliary-Pancreatic Surgery, Huadong Hospital Affliated to Fudan University
Brief Title: Predictors for Low Rates of Surgical Resection in Elderly Patients With Resectable Pancreatic Ductal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director of hospital, Fudan University
Other Study IDs: HuaDong Hosiptal of FUDAN
Record Dates: First submitted 2024-03-20; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pancreatic ductal adenocarcinoma; elderly; treatment abandonment; relative weight analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group of undergoing radical surgery: Elderly patients diagnosed with resectable PDAC underwent radical surgery.
- group of abandoning radical surgery: Elderly patients diagnosed with resectable PDAC abandoned radical surgery, the reasons of treatment abandonment included surgeons didn't recommend surgery for their elderly patients and patients chose to refuse surgery.
  Interventions: Other: potential predictors

INTERVENTIONS:
Other: potential predictors — Researchers want to investigate some important factors that influence elderly patients not to undergo radical surgery.
  Groups: group of abandoning radical surgery

SUMMARY:
More and more older adults are diagnosed with pancreatic ductal adenocarcinoma (PDAC), but the rate of surgical resection in patients with resectable tumour is still low. Clinical workers need to take more attention to oncologic care in this group. It's significant to explore potential predictors for impacting elderly patients chose to abandon surgical resection.

DETAILED DESCRIPTION:
The incidence of pancreatic ductal adenocarcinoma (PDAC) in the elderly has been on the rise, but the elderly were always neglected in clinical oncology care. Pancreatic ductal adenocarcinoma is a lethal disease, and the most effective treatment for curing it remains the radical resection. Unfortunately, there are many a study had reported that the rate of radical surgery of patients with PDAC has been low in the past decade. In order for more elderly pancreatic cancer patients to undergo surgical resection, investigators extracted the data of elderly patients with PDAC from SEER program and investigated predictive factors associated with surgical resection abandonment. In this study, investigators extracted data of patients older than 75 years diagnosed with T1-T3 stage PDAC to investigate rate of radical surgery. And researchers used Univariate and multivariate logistic regression model to explore potential factors associated with patients and surgeon chose to abandon surgical resection.

ELIGIBILITY:
Inclusion Criteria:

1. patients older than 75 years old and were diagnosed with pancreatic ductal adenocarcinoma by positive histology.
2. Patients were diagnosed with T1 through T3, M0 tumor based on criteria of TNM stage.

Exclusion Criteria:

1. Patients were diagnosed by death certificate.
2. Patients died before radical surgery.
3. Patients with important data missing, such as T-stage, surgical resection status, surgery procedures and complete survival time.

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Researchers included all elderly patients with T1-T3 stage PDAC recorded in SEER program, which would be candidates for undergoing radical surgery. Patients with metastatic disease were excluded. In addition, Investigators want to demonstrate survival benefit of radical surgery for elderly patients, so patients without complete survival time were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 5302 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
ORs of potential predictors | months from diagnosis to surgical resection, up to 12 months
  Univariate and multivariate logistic regression model were used to calculate ORs

SECONDARY OUTCOMES:
Overall survival (OS) | up to 132 months
  The date of definite diagnosis to death or last follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong Hospital affiliated to Fudan University, Shanghai, China